CLINICAL TRIAL: NCT05909605
Title: Non-invasive Measurements of Arterial Pulses and Blood Pressure Using a Novel Ultrasound Patch
Brief Title: Clinical Feasibility of a Conformal Ultrasound Blood Pressure Sensor
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheng Xu, Associate Professor, University of California, San Diego
Other Study IDs: 804119, 191474, 191527, 210799
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Feasibility Study; Medical Device
MeSH Terms: interventions — Sphygmomanometers; Vascular Access Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound blood pressure sensor
  Interventions: Device: sphygmomanometer; Device: Arterial Line

INTERVENTIONS:
Device: sphygmomanometer — Comparison to the ultrasound sensor
Device: Arterial Line — Comparison to the ultrasound sensor

SUMMARY:
Blood pressure (BP) monitoring is essential for managing cardiovascular diseases. Arterial line (A-line), the clinical gold standard for BP monitoring, is too invasive for routine measurements. The sphygmomanometer, on the other hand, is non-invasive but captures only discrete values. The recently introduced conformal ultrasound sensor oﬀers non-invasive and continuous monitoring of BP, which can potentially improve the quality of patient care, but its accuracy has yet to be thoroughly validated. Here the investigators are working to validate the accuracy of a redesigned ultrasound sensor with enhanced reliability in BP measurements at-home and in clinics even under different interventions.

ELIGIBILITY:
Inclusion Criteria:

* Are able to provide informed consent
* Have at least one arm

Exclusion Criteria:

* Active cardiac arrhythmias
* Any other unstable, active medical condition (i.e., cardiac arrythmia, uncontrolled diabetes, active heart failure, active liver failure)
* Currently pregnant (this will be confirmed with a urine pregnancy test in women of childbearing potential)
* Any large movements of the arms (e.g., chorea, dyskinesias, ballism), that in the investigators' opinion, would make it difficult to measure blood pressure using a standard blood pressure cuff
* Any active skin infection or wound on the arm that would interfere with the devices used to measure blood pressure
* Diagnosis of dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants without any severe cardiac anomalies
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Device comparison to standard monitoring (Sphygmomanometer) | 2 years
  Clinical feasibility of the calibration accuracy of the non-invasive ultrasound blood pressure sensor in comparison to a sphygmomanometer on 10 participants.
Device comparison to standard monitoring (A-line) | 2 years
  Clinical feasibility of the ultrasound blood pressure sensor for monitoring trend changes for continuous 12 hours of measurement in comparison to an arterial line in the Intensive Care Unit on 10 participants.
Device comparison to standard monitoring (A-line) | 3 years
  Clinical feasibility of the ultrasound blood pressure sensor in comparison to an arterial line in the catheterization laboratory on 40 participants.
Device comparison to standard monitoring (Sphygmomanometer) | 4 years
  Clinical feasibility of the device accuracy of the non-invasive ultrasound blood pressure sensor in comparison to a sphygmomanometer on 90 participants in consulting room on orthostatic hypotension participants.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No